CLINICAL TRIAL: NCT01414686
Title: Commercially-Available Interactive Video Games for Individuals With Chronic Mobility and Balance Deficits Post-Stroke
Brief Title: Virtual Environment Rehabilitation for Chronic Stroke
Acronym: VEHAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Stacy Fritz, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00001904
Record Dates: First submitted 2011-08-08; First posted 2011-08-11 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment Group (Experimental)
  Interventions: Other: Commercially-Available Interactive Video Games
- Delayed Treatment Group (No Intervention)

INTERVENTIONS:
Other: Commercially-Available Interactive Video Games — Two commercially available gaming platforms were used in this study, the Nintendo Wii and the Sony PS 2. The Wii games included "Wii Sports" and "Wii Fit"; PS games included the EyeToy "Play 2" and "Kinetic". Each of these games provides multiple mini games which pose different movement challenges, including dynamic balance, speed, accuracy, general mobility, and weight shifts.
  Game play was performed 1 hour/day, 4 days/ week, for a period of 5 weeks, totaling 20 hours.
  Other Names: Gaming; Nintendo Wii; Playstation; Stroke
  Arms: Immediate Treatment Group

SUMMARY:
More than half of individuals post-stroke have residual movement disabilities, including reduced mobility, balance, and increased risk of falling. There is a need for innovative, long-term and economically-feasible interventions for those with chronic stroke. Recently, a focus has been placed on the use of virtual reality and interactive gaming as a low cost and effective manner of treating movement disorders. Yet few studies have investigated interactive gaming platforms effect on balance following stroke. The proposed study is a randomized, single-blind, control group cross-over study for individuals with chronic stroke designed to examine an innovative therapeutic approach by investigating the effects of commercially-available gaming systems on balance, mobility and fear of falling in a sample of individuals with chronic motor deficits following stroke.

DETAILED DESCRIPTION:
Objective: To determine if playing active video games results in improved balance and motor performance.

Design: Randomized-matched, single-blind, control group cross-over study Setting: Laboratory Patients: Participants with chronic hemiparesis post-stroke were randomly assigned to a gaming group or normal activity control group.

Interventions: Gaming systems provided an interactive interface of real-time movement of either themselves or an avatar on the screen. Participants played games 1 hour/day, 4 days/week, for 5 weeks, totaling 20 hours of game-play. The intervention was strictly game-play without physical therapy. All games were played in standing position and trainers supervised to protect against loss of balance.

Measurements: Both groups were tested prior to and following the 5 weeks (post-test) and 3 months following the completion of the intervention/control. Outcome measures included: Fugl-Meyer Motor Exam, Single Leg Stance time, symmetrical weight bearing, Berg Balance Scale, Dynamic Gait Index, Timed Up and Go, Six Minute Walk, 3 Meter Walk, step length differential, and perception of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 6 months following stroke
* Ability to walk 10 feet with or without assistance
* 18 years of age or older
* Clinical presentation of unilateral hemiplegia post-stroke
* Ability to follow simple two-step instructions

Exclusion Criteria:

* Unable to ambulate 150 feet prior to stroke
* History of serious chronic obstructive pulmonary disease or oxygen dependence
* Severe weight bearing pain
* Lower-extremity amputation
* Non-healing ulcers on the lower extremity
* Renal dialysis or end stage liver disease
* Legal blindness or deafness or severe visual or hearing impairment
* A history of significant psychiatric illness defined by diagnosis of bipolar affective disorder, psychosis, or schizophrenia
* Life expectancy less than one year
* Severe arthritis or orthopaedic problems that limit passive ranges of motion of lower extremity: Knee flexion contracture of -10 degrees, Knee flexion ROM < 90 degrees, hip flexion contracture > 25 degrees, ankle plantar flexion contracture > 15 degrees
* History of deep venous thrombosis or pulmonary embolism within 6 months
* Uncontrollable diabetes: diabetic coma, frequent insulin reactions
* Severe hypertension with systolic > 200mmHg and diastolic > 110mmHg at rest
* Intracranial hemorrhage related to aneurysm rupture or an arteriovenous malformation (hemorrhagic infarctions will not be excluded)
* History of severe seizure disorder; other neurological conditions such as multiple sclerosis or Parkinson's Disease
* Pain that is scored greater than 5 out of 10 on a visual analog scale and limits daily activity
* Any health problems judged by their screening physician to put the client at significant risk of harm during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Balance (Berg Balance Scale) | change from pre to post and change from pre to follow-up (3 months)
  Do determine the influence of active gaming on balance in individuals with chronic stroke

SECONDARY OUTCOMES:
balance (Berg Balance Scale) | change from pre to post and change from pre to follow-up (3 months)
  Determine whether the Nintendo Wii games or the Sony PlayStation 2 EyeToy a) offers superior improvement of balance
balance (Berg Balance Scale) | post (5 weeks)
  Determine whether individuals with low or high fall risk show greater improvements in balance following participation in an interactive video game session.
Participant Perception | Post test (5 weeks)
  Determine whether the Nintendo Wii games or the Sony PlayStation 2 EyeToy offers superior participant perception of 1) enjoyability of the game, 2) feasibility for independent use of the game, and 3) improvement in perceived mobility as a result of the game.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy L Fritz, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina - Public Health Research Building, Columbia, South Carolina, United States

REFERENCES:
- See also: University of South Carolina Rehabilitation Lab Website — http://www.sph.sc.edu/dpt/dpt-rehab/vehab.htm